CLINICAL TRIAL: NCT04315233
Title: A Phase I/Ib Trial of the CDK4/6 Antagonist Ribociclib And The HDAC Inhibitor Belinostat In Patients With Metastatic Triple Negative Breast Cancer And Recurrent Ovarian Cancer With Response Prediction By Genomics (CHARGE)
Brief Title: Ribociclib&Belinostat In Patients w Metastatic Triple Neg Breast Cancer & Recurrent Ovarian Cancer w Response Prediction By Genomics
Acronym: CHARGE
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Novartis (Industry); Acrotech Biopharma (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCI130492
Record Dates: First submitted 2020-03-17; First posted 2020-03-19 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Metastatic Breast Cancer; Recurrent Ovarian Carcinoma
MeSH Terms: conditions — Breast Neoplasms; Ovarian Neoplasms | interventions — ribociclib; belinostat

STUDY DESIGN:
Intervention Model Description: modified 3+3 dose escalation followed by an expansion cohort at the identified Recommended Phase 2 Dose (RP2D). Dose escalation will be open to the enrollment of patients diagnosed with triple-negative breast cancer or ovarian cancer. However, dose expansion will only be open to the enrollment of patients diagnosed with triple-negative breast cancer
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1: Dose Escalation Cohort (Experimental): Ribociclib and belinostat will be given at escalating doses and on multiple administration schedules throughout the dose escalation component of the study. The MTD identified in the dose escalation component will be used to define the dose and administration schedule used in the dose expansion.
  Interventions: Drug: Ribociclib; Drug: Belinostat
- Cohort 2: Dose expansion cohort (Experimental): Participant will be enrolled in dose expansion cohort at the identified Recommended Phase 2 Dose (RP2D). Dose escalation will be open to the enrollment of patients diagnosed with triple-negative breast cancer or ovarian cancer. However, dose expansion will only be open to the enrollment of patients diagnosed with triple-negative breast cancer
  Interventions: Drug: Ribociclib; Drug: Belinostat

INTERVENTIONS:
Drug: Ribociclib — Ribociclib Dose Level 0 (starting dose) 200mg QD Dose Level 1A 400mg QD on Days 8-28 Dose Level 1B 200mg QD Dose Level 2 400mg QD on Days 8-28
Drug: Belinostat — Belinostat Dose Level 0 (starting dose) 600mg/m2 daily for 5 days Dose Level 1A 600mg/m2 daily for 5 days Dose Level 1B 1000mg/m2 daily for 5 days Dose Level 2 1000mg/m2 daily for 5 days
  *Administration on 5 consecutive days is preferred. Administration within 7 days allowed as needed to accommodate holidays and infusion schedules.

SUMMARY:
This is an open-label, multi-center, phase I study designed to assess the maximum tolerated dose of ribociclib and belinostat in combination. The trial will open with a dose escalation followed by an expansion cohort at the identified dose. Dose escalation will be open to the enrollment of patients diagnosed with triple-negative breast cancer or ovarian cancer. Dose expansion will only be open to patients diagnosed with triple-negative breast cancer.

DETAILED DESCRIPTION:
We hypothesize that ribociclib plus belinostat will be a well-tolerated and demonstrate activity in women with metastatic triple-negative breast or recurrent ovarian cancers.

This trial combines two targeted agents, a CDK inhibitor and a lysine deacetylase (DAC) inhibitor for use as the first targeted treatment for metastatic triple-negative breast cancer. This in itself would be a leap forward for women who currently endure sequential treatment with cytotoxic chemotherapies. However, we will also be using samples from this trial in NIH-funded research on clonal evolution and geographic heterogeneity in breast cancer. Blockade of CDK4/6 and of lysine deacetylases (DAC) are both promising treatments for breast cancer. DAC inhibitors have been shown to have single-agent activity against triple-negative breast cancer in vivo, possibly through decreasing EMT, decreasing migration, and decreasing metastasis [6, 7] CDK4/6 inhibitor monotherapy causes cell cycle arrest and tumor regression in triple-negative breast cancer models. [8, 9] However, neither approach has been successfully translated into clinical use as a monotherapy.

There are several lines of evidence demonstrating that inhibiting DAC increases the sensitivity of breast cancer to CDK4/6 inhibition. Recently, we showed that inhibitors of cell cycle progression, including CDKN1A, CDKN1C, CDKN2B, and CDKN2D, are increased by DAC inhibition in breast cancer cell lines, including triple-negative cell lines. [10] Others have shown cell cycle arrest by DAC inhibitors due to increases in p21 or decreases in CDK2 and cyclin A. [11-13] We also see an increase in RB1 expression in breast cancer cell lines. In the TCGA breast cancer analysis, RB1 was frequently down-regulated but not mutated or lost in triple-negative breast cancer. [14] Therefore, we hypothesized that DAC inhibition would increase the sensitivity of breast cancer to CDK4/6 inhibition. We first tested this hypothesis in a small panel of cell lines. We showed and published that all showed synergy between a CDK4/6 inhibitor (PD-0322991) and DAC inhibitors. [10] Since then, we have tested the combination of the DAC inhibitor vorinostat and the CDK4/6 inhibitor PD-322991 in a larger panel of cell lines and have shown at least additivity in most triple-negative cell lines. Indeed, it seems that those cancers least sensitive to CDK4/6 inhibition may benefit the most from co-treatment with a DAC inhibitor.

Recently, we investigated ribociclib and belinostat in six triple-negative breast cancer cell lines. All 6 cell lines showed growth inhibition with belinostat and panobinostat. Synergy was seen in four of the six cell lines at multiple doses.

We have also recently completed an analysis on a window of opportunity trial of the DAC inhibitor high-dose valproic acid, in breast cancer.[15] In that study, women were treated with valproic acid for one week before definitive therapy began. Fifty percent of women with triple-negative breast cancers had a significant decrease in Ki-67 with one week of valproic acid, providing proof of principle biologic activity of DAC inhibition in triple-negative breast cancer. (By contrast, no HER2 positive tumor had a decrease in Ki-67 with valproic acid treatment.) Given the genomic similarities between serous ovarian cancer and triple-negative breast cancer seen in the TCGA and pan-cancer analyses [16], we have chosen to include ovarian cancers in the dose-escalation component to increase accrual rate but not in the dose-expansion.

Neither CDK4/6 inhibition nor DAC inhibition have a well-defined predictive biomarker to determine which cancers will respond and which will not. Because of the complex genomic effects of inhibition of the 11 DACs and the multiple targets of DACs, including histones, p53, etc, it is unlikely that a single gene or protein alteration will predict sensitivity. We have published a method for predicting sensitivity to targeted drugs using genome-wide gene expression analysis. [17] After demonstrating proof of principle by accurately predicting sensitivity to vemurafenib, we developed a genomic biomarker for the DAC inhibitor valproic acid. We then validated that this biomarker predicted sensitivity in vitro and in vivo. In the window of opportunity discussed above, our genomic signature had an AUC of 0.66 for predicting decreased Ki-67 with one week of treatment with valproic acid. We will develop a similar multi-gene gene expression based biomarker for the combination of ribociclib and belinostat.

ELIGIBILITY:
Inclusion Criteria:

For dose escalation cohorts only:

- Pathologically confirmed breast cancer with the following features:

* Measurable disease by RECIST 1.1;
* ER and PR ≤ 1% by immunohistochemistry;
* Her-2/neu negative (0 or 1+ by immunohistochemistry OR not-amplified by CAP/ASCO standards);
* Metastatic or unresectable and locally advanced and not amenable to treatment with curative intent, in the opinion of the enrolling investigator.

OR --Pathologically confirmed serous ovarian cancer that is recurrent and is unresectable, in the opinion of the enrolling investigator.

For dose expansion cohort only:

- Pathologically confirmed breast cancer with the following features:

* Measurable disease by RECIST 1.1;
* ER and PR ≤ 1% by immunohistochemistry;
* Her-2/neu negative (0 or 1+ by immunohistochemistry OR not-amplified by CAP/ASCO standards);
* Metastatic or unresectable and locally advanced and not amenable to treatment with curative intent, in the opinion of the enrolling investigator.

For all patients:

* Age ≥ 18.
* ECOG performance Status ≤ 2.
* Able to swallow pills.
* Adequate organ function as defined as:

  * Hematologic:

    * ANC > 1,500/mm3
    * Platelets > 100,000/mm3
    * Hemoglobin > 9g/dL
  * Hepatic:

    * Serum bilirubin levels ≤1.5 mg/dL. Higher levels are acceptable if these can be attributed to active hemolysis or ineffective erythropoiesis. Bilirubin above 1.5mg/dL due to Gilbert's is still excluded.
    * Serum aspartate transaminase (AST) and serum alanine transaminase (ALT) ≤ 2.5 X upper limit of normal.
    * AST(SGOT)/ALT(SGPT) ≤ 5 × institutional ULN for patients with liver metastasis.
    * Alkaline phosphatase < 2.5 X upper limit of normal, unless bone metastasis is present in the absence of liver metastasis
  * Renal:

    * Serum creatinine levels ≤1.5 mg/dL
    * Patient must have the following laboratory values within normal limits or corrected to within normal limits with supplements before the first dose of study medication:

      * Potassium
      * Magnesium
      * Total Calcium (corrected for serum albumin)
  * Coagulation ---INR ≤1.5 (unless the patient is receiving anticoagulants and the INR is within the therapeutic range of intended use for that anticoagulant within 7 days prior to the first dose of study drug)
* Presence of ≥ 1 metastatic sites of disease that can be safely accessed for biopsy and patient willingness to undergo fresh tissue biopsies of up to 3 lesions. (Safely accessible means risk of mortality or major morbidity < 1.5%, such as core needle biopsy of breast, superficial lymph node, subcutaneous nodule, peripheral liver nodule, pleural nodule, omental nodule, etc. or per investigator discretion)
* Negative serum or urine pregnancy test at screening for women of childbearing potential.
* Agrees to continue use of approved birth control for at least 6 months after receiving the last dose of study drugs. See section 7.3 for list of approved birth control methods.
* Able to provide informed consent and have signed an approved consent form that conforms to federal and institutional guidelines.

Exclusion Criteria:

* Previous use of CDK 4/6 or HDAC inhibitors for cancer treatment
* Major surgery, radiotherapy, anticancer therapy, or investigational agents ≤ 4 weeks of treatment day 1 or ≤5 half-lives, whichever is shorter.
* Patients with new or progressive brain metastases (active brain metastases) or leptomeningeal disease unless determined by the treating physician that immediate CNS specific treatment is not required and is unlikely to be required during the first cycle of therapy.
* Medical condition that in the opinion of the enrolling investigator would require the use of valproic acid within ≤ 5 days of the first dose of belinostat or while on study.
* Active infection requiring systemic therapy.
* History of allergy or hypersensitivity to belinostat, ribociclib, or their binders.
* Uncontrolled arrhythmia, congestive heart failure or angina. Patients who have had a myocardial infarction, symptomatic pericarditis, or cardiac surgery should be at least 6 months from the event and free of active symptoms
* Known left ventricular ejection fraction < 50%. (Echocardiogram is not required for study entry)
* Clinically significant cardiac arrhythmias (e.g., ventricular tachycardia), complete left bundle branch block, high-grade AV block (e.g., bifascicular block, Mobitz type II and third degree AV block)
* Congenital long QT syndrome.
* Baseline QTcF>450 msec. The heart rate on the qualifying ECG must be between 50 and 90 BPM.
* Concurrent use of medication known to inhibit UGT1A1. Patients currently taking these medications must have discontinued ≥7 days prior to treatment day 1.
* Concurrent use of herbal supplements, unless approved by the prinicipal investigator. Patients currently taking herbal supplements must have discontinued ≥ 7 days prior to treatment day 1.
* Concurrent use of medication with a known risk of inducing Torsades de Pointes (on the known risk list of crediblemeds.org) that cannot be discontinued or switched to a different medication ≥ 7 days prior to starting the study drug.
* Unresolved diarrhea ≥ Grade 2, per CTCAE v5.0.
* Use of any of the following substances ≤ 7 days prior to the start of the treatment:

  * Known strong and moderate inducers or inhibitors of CYP3A4/5, including grapefruit, grapefruit hybrids, pomelos, star-fruit, and Seville oranges.
  * Medications that have a narrow therapeutic window and are predominantly metabolized through CYP3A4/5. Examples include certain benzodiazepines such as alprazolam and anti-seizure medications such as carbamazepine. Ultimately determination of drugs with a narrow therapeutic window is left to the discretion of the principal investigator.
* Patient is currently receiving warfarin or other coumarin derived anti-coagulant, for treatment, prophylaxis or otherwise.

  --Note: Therapy with heparin, low molecular weight heparin (LMWH), an oral factor Xa inhibitor, an oral direct thrombin inhibitor, or fondaparinux is allowed.
* Impaired GI function that may alter absorption of medicines, such as uncontrolled inflammatory bowel disease, uncontrolled vomiting, or major stomach or small bowel resection.
* Pregnant or breast feeding
* Women of child-bearing potential defined as all women physiologically capable of becoming pregnant or men whose female partner is of child-bearing potential, unless they are using highly effective methods of contraception during the study treatment and for 6 months after stopping the treatment. Highly effective contraception methods include:

  * Total abstinence (when this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception
  * Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy), total hysterectomy or tubal ligation at least 6 weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment
  * Male partner sterilization (at least 6 months prior to screening). For female patients on the study, the vasectomized male partner should be the sole partner for that patient and the success of the vasectomy must be medically confirmed as per local practice.
  * Placement of an intrauterine device (IUD).
  * Use of hormonal contraception plus a barrier contraceptive.
* Known HIV infection with a detectable viral load within 6 months of the anticipated start of treatment.

Note: Patients on effective anti-retroviral therapy with an undetectable viral load within 6 months of the anticipated start of treatment are eligible for this trial.

* Known chronic hepatitis B virus (HBV) or hepatitis C virus infection with a detectable viral load.

  --Note: Patients with an undetectable HBV viral load on appropriate suppressive therapy are eligible. Patients with an undetectable HCV viral load are eligible.
* Malignancy other than breast carcinoma or ovarian cancer (dose escalation) anticipated to need systemic treatment within 1 year in the opinion of the enrolling investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2021-05-03 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
MTD of ribociclib and belinostat combination | C1D1 to C2D1 (each cycle is 28 days)
  incidence of DLTs during the defined DLT period

SECONDARY OUTCOMES:
frequency and characterization of AEs and SAEs | 36 months
  safety of ribociclib and belinostat combination
Progression Free Survival (PFS) | 36 months
  assess efficacy
Objective Response Rate (ORR) | 36 months
  assess efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Theresa Werner, MD, Principal Investigator — Huntsman Cancer Institute
Locations (2):
- United States (2):
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Inova Schar Cancer Institute, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No